CLINICAL TRIAL: NCT03770091
Title: Impact of Theraworx Foam on Pain and Motion and Patient-Reported Outcomes in Thumb Arthritis
Brief Title: Impact of TheraWorx Foam on Symptom Relief in Thumb Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: John Fowler (Other)
Responsible Party: Sponsor-Investigator, John Fowler, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY18090019
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Results first posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Foam and Compression Wrap (Experimental): Patients will use Theraworx foam and a compression wrap
  Interventions: Drug: Theraworx
- Placebo Foam and Compression Wrap (Placebo Comparator): Patients will use placebo foam and a compression wrap
  Interventions: Drug: Placebo
- Foam alone (Experimental): Patients will use Theraworx foam without compression wrap
  Interventions: Drug: Theraworx

INTERVENTIONS:
Drug: Theraworx — Theraworx foam applied to skin and/or compression wrap
  Arms: Foam alone; Foam and Compression Wrap
Drug: Placebo — Placebo foam
  Arms: Placebo Foam and Compression Wrap

SUMMARY:
Thumb carpometacarpal osteoarthritis (CMC OA) affects up to 33% of people over the age of 40, which leads to inflammation, pain, and weakness of the CMC joint. Treatment modalities are both conservative and surgical with surgical options including osteotomy, bone excision, ligament reconstruction, and various prosthetic implants. The conservative treatment options, however, are limited to NSAIDs and bracing or steroid injections.

Advances in topical therapies have the potential to deliver focused treatment to the CMC joint. Novel treatment of inflammation can potentially reduce inflammation and pain associated with progressing osteoarthritis. Theraworx Relief is an FDA registered foam that has theoretical impact on inflammation reduction in human subjects treated with the topical foam.

DETAILED DESCRIPTION:
This pilot study seeks to investigate potential benefit in the use of Theraworx Foam in patients diagnosed with thumb CMC OA. Patients presenting to the upper extremity orthopedic surgery clinic for thumb/hand/wrist pain will be diagnosed by a Board Certified Hand Surgeon as per standard protocols. Patients who are recommended to follow a conservative treatment modality and are interested in participating in this study will be randomized into treatment or control groups. Both groups will undergo symptom assessment, strength testing, and range of motion testing prior to starting the standard conservative treatment of bracing. The treatment group will use the TheraWorx topical foam and the compression wrap nightly for 2 weeks for at least 6 hours per night. Control group will use a compression wrap for the same time period. Both groups will return at 1 and 2 weeks for repeat strength and range of motion testing and symptom assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Thumb CMC arthritis
2. greater than or equal to age 18
3. Interested in non-operative treatment of thumb arthritis

Exclusion Criteria:

1. Recent corticosteroid injection into the thumb joint
2. Non-English speaking
3. skin lesions or rashes on the thumb
4. current use of topical anti-inflammatory medications
5. concomitant thumb/wrist diagnoses that would impact the results (as determined by the PI)
6. known allergy to magnesium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John R Fowler, MD, Principal Investigator — Univ. of Pittsburgh Orthopaedic Surgery
Locations (3):
- United States (3):
  - Kaufmann Building, Pittsburgh, Pennsylvania
  - Montefiore Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Foam and Compression Wrap | Placebo Foam and Compression Wrap | Foam Alone
Started | 15 | 13 | 12
Completed | 15 | 13 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Foam and Compression Wrap | Placebo Foam and Compression Wrap | Foam Alone | Total
Number analyzed (Participants) | 15 | 13 | 12 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 8 | 26
  >=65 years | 5 | 5 | 4 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (10) | 60 (8) | 60 (9) | 60 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 11 | 38
  Male | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 1 | 5
  White | 13 | 11 | 11 | 35
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 13 | 12 | 40

OUTCOME MEASURES:

1. Primary Outcome: Numeric Pain Rating Scale
Description: patient rated pain on scale of 0-10 (0 no pain and 10 maximum pain). The mean score at 2 weeks is reported, not the change from baseline.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Foam and Compression Wrap | Placebo Foam and Compression Wrap | Foam Alone
Number analyzed (Participants) | 15 | 13 | 12
units on a scale | 1.7 (1.3) | 2.4 (1.5) | 3.2 (2.1)
Statistical Analysis 1: Comparison: Foam and Compression Wrap vs Placebo Foam and Compression Wrap vs Foam Alone; Test type: Superiority — ANOVA performed; p = 0.6, ANOVA

2. Primary Outcome: Disabilities of the Arm, Shoulder, and Hand (DASH) Score
Description: patient rated outcome score on scale of 0-100, with 0 being no disability and 100 complete disability, mean value at 2 weeks is reported
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Foam and Compression Wrap | Placebo Foam and Compression Wrap | Foam Alone
Number analyzed (Participants) | 15 | 13 | 12
score on a scale | 22.8 (10.9) | 35.9 (17.1) | 26.35 (12.5)
Statistical Analysis 1: Comparison: Foam and Compression Wrap vs Placebo Foam and Compression Wrap vs Foam Alone; Test type: Superiority; p = 0.59, ANOVA

3. Primary Outcome: Thumb Range of Motion
Description: This measures range of motion of the thumb in degrees from 0-90 degrees (0 degrees would be no motion and 90 degrees full motion), 2 week data is presented as a mean.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Foam and Compression Wrap | Placebo Foam and Compression Wrap | Foam Alone
Number analyzed (Participants) | 15 | 13 | 12
degrees | 70 (10) | 60 (12) | 70 (10)
Statistical Analysis 1: Comparison: Foam and Compression Wrap vs Placebo Foam and Compression Wrap vs Foam Alone; Test type: Superiority; p = 0.9, ANOVA

4. Primary Outcome: Grip Strength
Description: This measures grip strength in pounds (0 is no grip strength 150 is maximum grip strength), mean grip strength in pounds reported at 2 weeks
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Foam and Compression Wrap | Placebo Foam and Compression Wrap | Foam Alone
Number analyzed (Participants) | 15 | 13 | 12
pounds | 74 (9.6) | 67 (8.7) | 72 (9.4)
Statistical Analysis 1: Comparison: Foam and Compression Wrap vs Placebo Foam and Compression Wrap vs Foam Alone; Test type: Superiority; p = 0.45, ANCOVA

5. Primary Outcome: Pinch Strength
Description: This measures pinch strength in pounds (0 is no pinch strength and 40 is maximum pinch strength), mean pinch in pounds reported at 2 weeks
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Foam and Compression Wrap | Placebo Foam and Compression Wrap | Foam Alone
Number analyzed (Participants) | 15 | 13 | 12
pounds | 22.5 (10.5) | 29 (17.1) | 25 (14.7)
Statistical Analysis 1: Comparison: Foam and Compression Wrap vs Placebo Foam and Compression Wrap vs Foam Alone; Test type: Superiority; p = 0.5, ANOVA

ADVERSE EVENTS:
Time Frame: Collected information on reactions to foam or placebo over course of study (2 weeks)
Arm/Group | Foam and Compression Wrap | Placebo Foam and Compression Wrap | Foam Alone
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/15 | 0/13 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT03770091/Prot_SAP_001.pdf